CLINICAL TRIAL: NCT05642663
Title: Post-marketing, Observational Study of ALTUS Powered Stapler Used in Bariatric Surgery
Brief Title: Observational Study of ALTUS Powered Stapler Used in Bariatric Surgery
Status: Active, not recruiting | Type: Observational
Sponsor: Scitech Produtos Medicos Ltda (Industry)
Responsible Party: Sponsor
Other Study IDs: SCI-GE-001
Record Dates: First submitted 2022-11-18; First posted 2022-12-08 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-09

CONDITIONS: Obesity
Keywords: Stapler; ALTUS; Bariatric surgery
MeSH Terms: conditions — Obesity | interventions — Surgical Staplers

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Treated patients: Patients with grade II (with one or more associated comorbidities) and grade III obesity who went through sleeve, bypass and revisional bariatric surgery procedure with the use of Altus Powered Stapler
  Interventions: Device: Stapler

INTERVENTIONS:
Device: Stapler — Stapling performed with ALTUS Powered Stapler

SUMMARY:
Post-marketing, observational study to evaluate the safety and performance of the ALTUS Powered Stapler in bariatric surgery of "real-world" patients.

DETAILED DESCRIPTION:
Up to 300 patients who underwent sleeve, bypass or revisional bariatric surgery with the use of Altus Powered Stapler will be included in the study. The stapler should be used according to the Instructions for Use and according to the local practice.

The Altus Powered Stapler is used in open or laparoscopic surgeries and simultaneously cuts and staples soft tissues. In order to avoid great physical efforts by the physician and ensure excellent tissue suturing, the cutting and stapling mechanism is driven by the 12-volt battery that comes with the stapler.

Patients will be followed by 7, 30 and 90 days and 12 months after the procedure, as per the research center's standard routine.

ELIGIBILITY:
Inclusion Criteria:

* Patients with grade II obesity (BMI ≥ 35 kg/m^2) with one or more associated comorbidities;
* Patients with grade III obesity (BMI ≥ 40 kg/m^2) regardless of associated diseases;
* Patients who underwent sleeve, bypass and revisional bariatric surgery procedure with use of the Altus Powered Stapler;
* The patient must sign and date the informed consent form during a routine follow-up visit, authorizing the use of their surgery data and contact for follow-up.

Exclusion Criteria:

* Impossibility of collecting data related to the surgical procedure
* Impossibility of contact with the patient to obtain the informed consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults (18 years or older), who underwent bariatric surgery with the use of Altus Powered Stapler
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-05-31 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Safety - Conversion to open surgery | Intraoperative
  Number of conversions to open surgery during the index procedure
Safety - Number of reinterventions | Up to 1 week
  Number of reinterventions within 1 week after the procedure
Safety - Postoperative anastomotic leaking and intraluminal/intraperitoneal bleeding | 30 days
  Presence of complications of anastomotic leaking and intraluminal/intraperitoneal bleeding within 30 days after procedure
Safety- Fistula formation | 30 days
  Presence of fistula within 30 days after procedure
Safety - Stenosis | 90 days
  Detection of stenosis within 90 days after procedure
Performance - Procedure Success | Intraoperative
  Defined by completion of technique with the device for its intended use
Performance - Cicatrization of staple line | 90 days
  The absence of oozing/bleeding at the staple line

SECONDARY OUTCOMES:
Post-operative change in weight | 12 months
  Defined by preoperative weight (kg) minus postoperative weight (kg) divided by ideal body weight (kg) at the end of 12 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital IGESP, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No